CLINICAL TRIAL: NCT00120081
Title: Phase 1, Single-Center, Double-Blind, Placebo-Controlled, Randomized, Dose-Escalation Study to Compare the Safety, Tolerability, and Immunogenicity of Three Intramuscular Administrations of Na-ASP-2 Hookworm Vaccine in Healthy Adults Without Evidence of Hookworm Infection
Brief Title: Study of Na-ASP-2 Human Hookworm Vaccine in Healthy Adults Without Evidence of Hookworm Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: SVI-04-01
Record Dates: First submitted 2005-07-07; First posted 2005-07-15 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hookworm Infection
Keywords: Vaccine; Hookworm; Phase 1; Human Hookworm Infection; Na-ASP-2
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose (Experimental): 10 mcg Na-ASP-2/Alhydrogel
  Interventions: Biological: Na-ASP-2/Alhydrogel Hookworm Vaccine
- Medium dose (Experimental): 50 mcg Na-ASP-2/Alhydrogel
  Interventions: Biological: Na-ASP-2/Alhydrogel Hookworm Vaccine
- High dose (Experimental): 100 mcg Na-ASP-2/Alhydrogel
  Interventions: Biological: Na-ASP-2/Alhydrogel Hookworm Vaccine
- Saline placebo (Placebo Comparator): Saline placebo
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: Na-ASP-2/Alhydrogel Hookworm Vaccine — The recombinant hookworm protein Na-ASP-2 formulated on aluminum hydroxide adjuvant (Alhydrogel), in one of three dose concentrations, compared to a saline placebo control.
  Arms: High dose; Low dose; Medium dose
Biological: Saline placebo — Inactive saline placebo control
  Arms: Saline placebo

SUMMARY:
The primary objective of this clinical trial is to determine the safety and tolerability of the Na-ASP-2 Hookworm Vaccine in healthy subjects following the administration of 3 intramuscular (IM) injections of the vaccine over 16 weeks using 3 different doses. The secondary objective is to make a preliminary evaluation of the immunogenicity of each of the 3 doses of the vaccine in healthy volunteers.

DETAILED DESCRIPTION:
There is an urgent need for new tools to control human hookworm infection and to reduce its burden of disease in developing countries. This is especially true for children and women of reproductive age who represent populations that are highly vulnerable to the effects of hookworm disease. Up to 65,000 deaths annually have been attributed to human hookworm infection. However, the mortality estimates of hookworm pale in comparison to global disease burden estimates.

The primary approach to hookworm control worldwide has been the frequent and periodic use of benzimidazole anthelminthics for school-age children. However, school-based anthelminthic chemotherapy programs miss populations highly vulnerable to hookworm, including adolescent and adult women. In addition, high rates of hookworm re-infection occur within 4-12 months following anthelminthic chemotherapy, and there is evidence for diminished efficacy of benzimidazoles with frequent and periodic use, possibly because of emerging drug resistance. These concerns have prompted interest in developing alternative tools for hookworm control. Vaccination to prevent high intensity hookworm infection would alleviate the public health deficiencies of drug treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18 to 45 years of age.
* Signed informed consent.
* History, physical exam, and laboratory tests indicating good general health obtained prior to the first injection.
* All females must have a negative pregnancy test (FDA-approved test for β human chorionic gonadotropin [β-HCG]) on the day of the first injection.
* Serologic tests for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) are negative at screening.
* All subjects must agree to use an acceptable method of birth control from the start of screening until 2 weeks after the third injection. Acceptable methods for female subjects include hormonal contraceptives, intrauterine device (IUD), diaphragm with spermicide, condoms, abstinence, surgically sterile (hysterectomy), and surgically sterile partner. Acceptable methods for male subjects include surgical sterilization, condoms, partner who uses an acceptable method of birth control, and abstinence.

Exclusion Criteria:

* Any history of anaphylaxis or allergy to vaccine components or allergy to insect stings, including bee stings.
* A past or current history of hookworm infection.
* BMI < 18.0 or > 30.0.
* Recent (< 72 hours) history of febrile illness at the time of vaccination (temperature > 99.6°F or equivalent).
* Received any immune globulin or blood product 3 months prior to injection or scheduled within 4 weeks thereafter.
* Had vaccination with a live virus vaccine within 4 weeks before receipt of the vaccine or scheduled within 4 weeks thereafter.
* Had vaccination with a killed vaccine, or allergy treatment with antigen injections within 14 days of initial study injection.
* Received an investigational agent within 4 weeks of initial study injection.
* Known or suspected impairment of immunologic function including, but not limited to clinically significant liver disease, diabetes mellitus, moderate to severe kidney impairment (creatinine > 1.5), any history of malignancy (except squamous cell or basal cell skin cancer), HIV infection or autoimmune diseases, or concomitant immunosuppressive medication such as glucocorticosteroids.
* A history of essential hypertension, gastrointestinal abnormalities such as peptic ulcer disease, cardiac (ECG abnormalities), pulmonary, hepatic, renal, pancreatic, or neurologic disease.
* Taken prescription medications with the exception of subjects on a stable regimen (> 30 days) of: (1) hormone replacement therapy, (2) use of nasal steroids, (3) topical therapy, (4) certain classes of antidepressants (i.e., selective serotonin re-uptake inhibitors), (5) oral contraceptives, (6) nonsteroidal anti-inflammatory agents, or (7) antihistamines or decongestants for seasonal allergies taken as needed.
* Contraindication to IM injection such as anti-coagulant therapy or thrombocytopenia.
* Pregnant, nursing, or expecting to conceive during the study.
* Any history of chronic alcohol or drug abuse or current treatment with any known prescribed or over-the-counter supplements that may be hepatotoxins.
* Any subject who, in the Investigator's opinion, will be unable to adhere to protocol requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of three different doses of the Na-ASP-2 hookworm vaccine in healthy volunteers | For the duration of the study

SECONDARY OUTCOMES:
To determine the immunogenicity, both humoral and cellular, of the vaccine at specified time points following vaccination | 2, 8, 10, 16, 18, 24, and 48 weeks after the first injection

CONTACTS AND LOCATIONS:
Overall Officials: Gary Simon, M.D., Ph.D, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Bethony JM, Simon G, Diemert DJ, Parenti D, Desrosiers A, Schuck S, Fujiwara R, Santiago H, Hotez PJ. Randomized, placebo-controlled, double-blind trial of the Na-ASP-2 hookworm vaccine in unexposed adults. Vaccine. 2008 May 2;26(19):2408-17. doi: 10.1016/j.vaccine.2008.02.049. Epub 2008 Mar 11. PMID 18396361
- See also: Sponsor's Web page — http://www.sabin.org